CLINICAL TRIAL: NCT03335553
Title: Randomized, Double-Blind, Placebo-Controlled Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-986235 in Healthy Subjects
Brief Title: A Study of Experimental Medication BMS-986235 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV018-001
Record Dates: First submitted 2017-11-06; First posted 2017-11-07 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Mediators of Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single ascending dose (SAD): BMS-986235 or Placebo (Experimental): BMS-986235 or Placebo oral dose
  Interventions: Drug: BMS-986235; Other: Placebo
- Multiple ascending dose (MAD): BMS-986235 or Placebo (Experimental): BMS-986235 or Placebo oral dose
  Interventions: Drug: BMS-986235; Other: Placebo

INTERVENTIONS:
Drug: BMS-986235 — Specified dose on specified days
Other: Placebo — Specified dose on specified days

SUMMARY:
This is a study of experimental medication BMS-986235 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be normal healthy volunteers as determined by no clinically significant deviations in medical history, physical examination, ECGs, vital signs, and clinical laboratory determinations
* Patients must have a body mass index (BMI) of 18 - 30 mg/kg2, inclusive

Exclusion Criteria:

* Patients that are pregnant
* Patient with any significant acute or chronic medical illness
* Patient with a current or recent (within 3 months of study treatment administration) gastrointestinal disease that could affect absorption
* Patient with any surgery within 12 weeks of study treatment administration
* Patient with any gastrointestinal surgery that could impact upon the absorption of study drug
* Patient who donated blood to a blood bank or in a clinical study (except a screening visit) within 12 weeks of study drug administration (within 2 weeks for plasma only)
* Patient who received a blood transfusion within 12 weeks of study drug administration

Other protocol defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse events (SAE) | Approximately 30 days
Number of deaths | Approximately 30 days
Number of adverse events (AE) leading to study discontinuation | Approximately 30 days
Number of patients with clinically significant changes in ECG parameters, as defined by the investigator | Approximately 30 days
Number of patients with potentially clinically significant changes in vital signs | Approximately 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, Anaheim, California
  - PRA Health Sciences, Salt Lake City, Utah

REFERENCES:
- [Derived] Singh J, Jackson KL, Fang H, Gumanti A, Claridge B, Tang FS, Kiriazis H, Salimova E, Parker AM, Nowell C, Woodman OL, Greening DW, Ritchie RH, Head GA, Qin CX. Novel formylpeptide receptor 1/2 agonist limits hypertension-induced cardiovascular damage. Cardiovasc Res. 2024 Sep 21;120(11):1336-1350. doi: 10.1093/cvr/cvae103. PMID 38879891
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm